CLINICAL TRIAL: NCT00195494
Title: A 24-Month,Randomized,Double-Blind,Two-Period Study to Evaluate the Efficacy and Safety of the Combination of Etanercept and Methotrexate and Methotrexate Alone in Subjects With Early Rheumatoid Arthritis
Brief Title: Study Comparing Etanercept and Methotrexate vs. Methotrexate Alone in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0881A-101548
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1a (Active Comparator): Etanercept + Methorexate for Period 1 (first 12 months) and Period 2 (Second 12 months)
  Interventions: Drug: Etanercept; Drug: Methotrexate
- 1b (Active Comparator): Etanercept + Methotrexate for Period 1 (First 12 months) and Etanercept alone for Period 2 (Second 12 months)
  Interventions: Drug: Etanercept; Drug: Methotrexate; Drug: Placebo
- 2a (Active Comparator): Methotrexate alone in Period 1 (First 12 months) and etanercept + Methotrexate in Period 2 (Second 12 months)
  Interventions: Drug: Etanercept; Drug: Methotrexate; Drug: Placebo
- 2b (Active Comparator): Methotrexate alone in Period 1 (First 12 months) and Methotrexate alone in Period 2 (Second 12 months)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Etanercept — Group 1a: Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 1 & 2
  Group 1b: Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 1 then Etanercept 50 mg SC injections weekly + Placebo weekly for Period 2
  Group 2a: Oral Methotrexate weekly + Placebo for Period 1, then Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 2
  Arms: 1a; 1b; 2a
Drug: Methotrexate — Group 1a: Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 1 & 2
  Group 1b: Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 1 then Etanercept 50 mg SC injections weekly + Placebo weekly for Period 2
  Group 2a: Oral Methotrexate weekly + Placebo for Period 1, then Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 2
  Group 2b: Oral Methotrexate weekly for both Periods 1 and 2
Drug: Placebo — Group 1b: Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 1 then Etanercept 50 mg SC injections weekly + Placebo weekly for Period 2
  Group 2a: Oral Methotrexate weekly + Placebo for Period 1, then Etanercept 50 mg SC injections weekly + oral Methotrexate weekly for Period 2
  Arms: 1b; 2a

SUMMARY:
To compare the effects of the combination of ETN and MTX to MTX alone on radiographic change and clinical disease activity in subjects with early RA over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Satisfies the 1987 ACR Revised Criteria for Rheumatoid Arthritis
* Has RA greater than or equal to 3 months and less than or equal to 2 years

Exclusion Criteria:

* Received any previous treatment with MTX
* Received any previous treatment with ETN or other tumour necrosis factor antagonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Denver, Colorado, United States

REFERENCES:
- [Derived] Fleischmann RM, van der Heijde D, Gardiner PV, Szumski A, Marshall L, Bananis E. DAS28-CRP and DAS28-ESR cut-offs for high disease activity in rheumatoid arthritis are not interchangeable. RMD Open. 2017 Jan 30;3(1):e000382. doi: 10.1136/rmdopen-2016-000382. eCollection 2017. PMID 28255449
- [Derived] Gallo G, Brock F, Kerkmann U, Kola B, Huizinga TW. Efficacy of etanercept in combination with methotrexate in moderate-to-severe rheumatoid arthritis is not dependent on methotrexate dosage. RMD Open. 2016 Apr 21;2(1):e000186. doi: 10.1136/rmdopen-2015-000186. eCollection 2016. PMID 27175292
- [Derived] Zhang W, Sun H, Emery P, Sato R, Singh A, Freundlich B, Anis AH. Does achieving clinical response prevent work stoppage or work absence among employed patients with early rheumatoid arthritis? Rheumatology (Oxford). 2012 Feb;51(2):270-4. doi: 10.1093/rheumatology/ker189. Epub 2011 Jun 29. PMID 21719418
- [Derived] Emery P, Breedveld FC, Hall S, Durez P, Chang DJ, Robertson D, Singh A, Pedersen RD, Koenig AS, Freundlich B. Comparison of methotrexate monotherapy with a combination of methotrexate and etanercept in active, early, moderate to severe rheumatoid arthritis (COMET): a randomised, double-blind, parallel treatment trial. Lancet. 2008 Aug 2;372(9636):375-82. doi: 10.1016/S0140-6736(08)61000-4. Epub 2008 Jul 16. PMID 18635256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited worldwide from November 2004 to February 2006.
Pre-assignment Details: Participants were randomly assigned equally to 1 of 4 blinded treatment groups: Group (G) 1a received the combination of etanercept (E) and methotrexate (M) in year Y1 and Y2. G1b received the combination of E and M in Y1 and E alone in Y2. G2a received M alone in Y1 and the combination of E and M in Y2. G2b received M alone in Y1 and Y2.
Groups:
- Year 1 E+M / Year 2 E+M: Following a blinded transition from year one- Etanercept injection- two injections 25 mg weekly (given at the same time at different sites)+ oral Methotrexate capsules weekly (same day as injection).
  Dose consistent with the ending dose at year one (usually 20 mgs). No reduction of MTX dose is permitted in year two.
- Year 1 M / Year 2 E+M: Following a blinded transition from year one- Etanercept two injections 25 mg weekly (given at the same time at different sites) + oral Methotrexate capsules weekly (same day as injection).
  Dose consistent with the ending dose at year one (usually 20 mgs). No reduction of MTX dose is permitted in year two.
- Year 1 E+M / Year 2 E: Following a blinded transition from year one-Etanercept two injections 25 mg weekly (given at the same time at different sites).
- Year 1 M / Year 2 M: Following a blinded transition from year one- Methotrexate dose consistent with the ending dose of year one (usually 20 mgs).
  No reduction of MTX dose is permitted in year two.
- Year 1 M+Placebo: Oral Methotrexate capsules once weekly + two injections of placebo given at the same time at different sites.
  MTX dose is a forced titration from 7.5mg (3 capsules) to 20 mg weekly (8 capsules) by week 8.
- Year 1 E+M: Etanercept injection- two injections 25 mg weekly (given at the same time at different sites) + oral Methotrexate capsules weekly (same day as injection).
  MTX dose is a forced titration from 7.5mg (3 capsules) to 20 mg weekly (8 capsules) by week 8.
Period: Year 1
Arm/Group | Year 1 E+M / Year 2 E+M | Year 1 M / Year 2 E+M | Year 1 E+M / Year 2 E | Year 1 M / Year 2 M | Year 1 M+Placebo | Year 1 E+M
Started | 0 | 0 | 0 | 0 | 268 | 274
Completed | 0 | 0 | 0 | 0 | 189 | 221
Not Completed | 0 | 0 | 0 | 0 | 79 | 53
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 34 | 27
Not completed — System Toxicity | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 24 | 9
Not completed — Compliance | 0 | 0 | 0 | 0 | 5 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Missed >4 consecutive doses | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 8 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1
Period: Year 2
Arm/Group | Year 1 E+M / Year 2 E+M | Year 1 M / Year 2 E+M | Year 1 E+M / Year 2 E | Year 1 M / Year 2 M | Year 1 M+Placebo | Year 1 E+M
Started | 111 (A patient with Year 1 termination had taken drug briefly during Year 2 and thus counted in the data.) | 90 | 111 (A patient with Year 1 termination had taken drug briefly during Year 2 and thus counted in the data.) | 99 | 0 | 0
Completed | 104 | 74 | 93 | 76 | 0 | 0
Not Completed | 7 | 16 | 18 | 23 | 0 | 0
Not completed — Adverse Event | 3 | 7 | 5 | 9 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 7 | 7 | 0 | 0
Not completed — Compliance | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Missed >4 consecutive doses | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 4 | 3 | 0 | 0
Not completed — System toxicity | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Year 1 M+Placebo | Year 1 E+M | Total
Number analyzed (Participants) | 268 | 274 | 542
Age Continuous [Median (Full Range); unit: years] — Year 1 Overall Number of Baseline Participants is 542
  years | 51.50 [20.00 to 84.00] | 52.50 [18.00 to 82.00] | 52.00 [18.00 to 84.00]
Sex: Female, Male [Count of Participants; unit: Participants] — Year 1 participants collected from Arms M and E+M equal the stated overall participant population of 542. 411 of those participants were then entered into Year 2 Arms E+M/E+M, M/M+E, E+M/E, M/M. This measure provides the gender population for Year 1 only in order to accurately reflect the overall baseline population of 542.
  Participants
    Female | 194 | 204 | 398
    Male | 74 | 70 | 144

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Achieving Remission As Measured by a Disease Activity Score for 28 Joints (DAS 28) < 2.6.
Description: Effects of the combination of etanercept and methotrexate to methotrexate alone on clinical disease activity. DAS28 scale 0 - 10, 3.2 or lower showing controlled disease while 5.1 implies active disease.
Time Frame: 12 months
Population: The analysis population is the modified intent to treat participants from year 1, treatment arms M and E+M.
Measure: Number; unit: participants
Groups:
- Year 1 M: Oral methotrexate capsules 7.5mg weekly and etanercept placebo at the same day and time.
- Year 1 E+M: etanercept injection 50mg once weekly and oral methotrexate capsules 7.5 mg once weekly at the same time
Arm/Group | Year 1 M | Year 1 E+M
Number analyzed (Participants) | 263 | 265
participants | 73 | 132
Statistical Analysis 1: Comparison: Year 1 M vs Year 1 E+M; Test type: Superiority or Other; p < 0.001, Fisher Exact; Risk Difference (RD) = 22.0 — E+M (49.8%) - M (27.8%) creates the risk difference estimated value

2. Primary Outcome: Year 1 Participants Having an Annualized Modified Total Sharp Score (mTSS) < 0.5.
Description: The (van der Heijde) modified total Sharp score (mTSS) is the sum of scores for erosions (range 0-280) and joint space narrowings (range 0-168) and thus has a total range of (0 - 448 ), where zero is the best score , indicating no damage.
Time Frame: 12 months
Population: The analysis population is the modified intent to treat participants from year 1, treatment arms M and E+M.
Measure: Number; unit: participants
Arm/Group | Year 1 M | Year 1 E+M
Number analyzed (Participants) | 230 | 246
participants | 135 | 196
Statistical Analysis 1: Comparison: Year 1 M vs Year 1 E+M; Test type: Superiority or Other; p < 0.001, Fisher Exact; Risk Difference (RD) = 21.0 — E+M (79.7%) - M (58.7%) creates the risk difference estimated value

3. Secondary Outcome: Safety Measured by Number of Participants Reporting a Serious Adverse Event That Led to Death
Description: Safety report for entire trial where participants reported a serious adverse event that led to death.
Time Frame: 12 and 24 months
Population: The analysis population is the modified intent to treat for year 1 (542 overall baseline participants) and year 2 (411 overall baseline participants).
Measure: Number; unit: participants
Groups:
- Year 2 E+M / E+M: Following a blinded transition from year one- Etanercept injection- two injections 25 mg weekly (given at the same time at different sites)+ oral Methotrexate capsules weekly (same day as injection).
  Dose consistent with the ending dose at year one (usually 20 mgs). No reduction of MTX dose is permitted in year two.
- Year 2 M / E+M: Following a blinded transition from year one- Etanercept two injections 25 mg weekly (given at the same time at different sites) + oral Methotrexate capsules weekly (same day as injection).
  Dose consistent with the ending dose at year one (usually 20 mgs). No reduction of MTX dose is permitted in year two.
- Year 2 E+M / E: Following a blinded transition from year one-Etanercept two injections 25 mg weekly (given at the same time at different sites).
- Year 2 M / M: Following a blinded transition from year one- MTX dose consistent with the ending dose of year one (usually 20 mgs).
  No reduction of MTX dose is permitted in year two.
Arm/Group | Year 2 E+M / E+M | Year 2 M / E+M | Year 2 E+M / E | Year 2 M / M | Year 1 M+Placebo | Year 1 E+M
Number analyzed (Participants) | 111 | 90 | 111 | 99 | 268 | 274
participants | 0 | 0 | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Year 1 E+M / Year 2 E+M | Year 1 M / Year 2 E+M | Year 1 E+M / Year 2 E | Year 1 M / Year 2 M | Year 1 M+Placebo | Year 1 E+M
Serious Adverse Events (participants affected / at risk) | 8 | 11 | 10 | 12 | 34 | 33
Other Adverse Events (participants affected / at risk) | 91 | 71 | 89 | 79 | 241 | 246
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Year 1 E+M / Year 2 E+M | Year 1 M / Year 2 E+M | Year 1 E+M / Year 2 E | Year 1 M / Year 2 M | Year 1 M+Placebo | Year 1 E+M
Angina unstable (Cardiac disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Arrhythmia (Cardiac disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Aterial fibrillation (Cardiac disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 1/268 | 0/274
Myocardial infarction (Cardiac disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 1/268 | 0/274
Pericarditis (Cardiac disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Ventricular tachycardia (Cardiac disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Vertigo (Ear and labyrinth disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Photophobia (Eye disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Appendicitis perforated (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Gastritis (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 1/274
General gastrointestinal disorder (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 1/268 | 0/274
Mechanical ileus (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Vomiting (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Chest pain (General disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 1/274
General physical health deterioration (General disorders) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 1/274
Cholelithiasis (Hepatobiliary disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 2/274
Gallbladder disorder (Hepatobiliary disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Acute sinusitis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 1/99 | 1/268 | 0/274
Bronchitis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Chronic sinusitis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Diverticulitis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Gastroenteritis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Herpes zoster (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Lung infection (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Lyme disease (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Nasopharyngitis (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Pneumonia (Infections and infestations) | 0/111 | 1/90 | 0/111 | 1/99 | 1/268 | 1/274
Septic athritis staphylococcal (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Skin infection (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Streptococcal infection (Infections and infestations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Accidental overdose (Injury, poisoning and procedural complications) | 2/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Joint injury (Injury, poisoning and procedural complications) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Overdose (Injury, poisoning and procedural complications) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Pelvic fracture (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Procedural pain (Injury, poisoning and procedural complications) | 0/111 | 1/90 | 0/111 | 0/99 | 1/268 | 0/274
Radius fracture (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Spinal fracture (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 1/111 | 0/99 | 1/268 | 0/274
Blood alkaline phosphatase increased (Investigations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Hepatic enzyme increased (Investigations) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Transaminases increased (Investigations) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Diabetes mellitus (Metabolism and nutrition disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Hyponatraemia (Metabolism and nutrition disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Arthritis (Musculoskeletal and connective tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Intervetebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 2/274
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 2/268 | 0/274
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 5/268 | 2/274
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 1/111 | 1/99 | 1/268 | 0/274
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 0/99 | 3/268 | 0/274
Chronic lymphocytic leukamia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 1/274
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Cerebral haemorrhage (Nervous system disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Headache (Nervous system disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Paraesthesia (Nervous system disorders) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 1/274
Syncope (Nervous system disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Syncope vasovagal (Nervous system disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Anxiety (Psychiatric disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Sleep disorder (Psychiatric disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Renal failure (Renal and urinary disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Urinary retention (Renal and urinary disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 2/274
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Hip arthroplasty (Surgical and medical procedures) | 0/111 | 0/90 | 0/111 | 0/99 | 2/268 | 0/274
Hospitalisation (Surgical and medical procedures) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Deep vein thrombosis (Vascular disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Infarction (Vascular disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 0/268 | 1/274
Ischaemia (Vascular disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 1/268 | 0/274
Aortic valve stenosis (Cardiac disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Atrio ventricular block (Cardiac disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Mitral valve incompetence (Cardiac disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Abdominal pain upper (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Inguinal hernia (Gastrointestinal disorders) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Systemic inflammatory response system (General disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Bursitis infected staphylococcal (Infections and infestations) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 0/274
Pneumonia streptococcal (Infections and infestations) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Tonsillitis (Infections and infestations) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Concussion (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Device failure (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Fall (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Ligament injury (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Skull fractured base (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Arthropathy (Musculoskeletal and connective tissue disorders) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 0/274
Spondylolisthesis acquired (Musculoskeletal and connective tissue disorders) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 0/274
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Malignant melanoma of sights other than skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Cerebellar infarction (Nervous system disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Cerebral infarction (Nervous system disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Cerebrovascular accident (Nervous system disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Hydrocephalus (Nervous system disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Sciatica (Nervous system disorders) | 0/111 | 1/90 | 1/111 | 0/99 | 0/268 | 0/274
Confusional state (Psychiatric disorders) | 0/111 | 1/90 | 0/111 | 0/99 | 0/268 | 0/274
Renal and urinary disorders (Psychiatric disorders) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 0/274
Renal colic (Psychiatric disorders) | 1/111 | 0/90 | 0/111 | 0/99 | 0/268 | 0/274
Testicular torsion (Reproductive system and breast disorders) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Vaginal prolapse (Reproductive system and breast disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/111 | 1/90 | 0/111 | 1/99 | 0/268 | 0/274
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Cholecystectomy (Surgical and medical procedures) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
Haemorrhoid operation (Surgical and medical procedures) | 0/111 | 0/90 | 1/111 | 0/99 | 0/268 | 0/274
Aneurysm (Vascular disorders) | 0/111 | 0/90 | 0/111 | 1/99 | 0/268 | 0/274
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Year 1 E+M / Year 2 E+M | Year 1 M / Year 2 E+M | Year 1 E+M / Year 2 E | Year 1 M / Year 2 M | Year 1 M+Placebo | Year 1 E+M
Blood and lymphatic (Blood and lymphatic system disorders) | 6/111 | 2/90 | 2/111 | 4/99 | 4/268 | 20/274
Cardiac disorders (Cardiac disorders) | 0/111 | 5/90 | 3/111 | 1/99 | 14/268 | 14/274
Ear and labyrinth (Ear and labyrinth disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 16/268 | 11/274
Eye (Eye disorders) | 5/111 | 4/90 | 5/111 | 7/99 | 20/268 | 28/274
Abdominal pain upper (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 27/268 | 23/274
Diarhhea (Gastrointestinal disorders) | 4/111 | 2/90 | 6/111 | 7/99 | 20/268 | 24/274
Nausea (Gastrointestinal disorders) | 8/111 | 8/90 | 4/111 | 8/99 | 48/268 | 53/274
Vomiting (Gastrointestinal disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 18/268 | 11/274
Administration site conditions (General disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 50/268 | 67/274
Nasopharyngitis (Infections and infestations) | 10/111 | 10/90 | 10/111 | 13/99 | 42/268 | 44/274
Upper respiratory tract infections (Infections and infestations) | 6/111 | 8/90 | 5/111 | 9/99 | 19/268 | 18/274
Urinary tract infections (Infections and infestations) | 0/111 | 2/90 | 6/111 | 4/99 | 10/268 | 17/274
Post procedural nausea (Injury, poisoning and procedural complications) | 0/111 | 0/90 | 0/111 | 0/99 | 23/268 | 18/274
Investigations (Investigations) | 0/111 | 0/90 | 0/111 | 0/99 | 50/268 | 49/274
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6/111 | 6/90 | 4/111 | 15/99 | 36/268 | 13/274
Headache (Nervous system disorders) | 8/111 | 4/90 | 6/111 | 4/99 | 20/268 | 29/274
Psychiatric (Psychiatric disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 23/268 | 28/274
Renal and urinary (Renal and urinary disorders) | 8/111 | 5/90 | 2/111 | 5/99 | 19/268 | 21/274
Cough (Respiratory, thoracic and mediastinal disorders) | 7/111 | 2/90 | 8/111 | 6/99 | 26/268 | 23/274
Alopecia (Skin and subcutaneous tissue disorders) | 0/111 | 0/90 | 0/111 | 0/99 | 8/268 | 15/274
Rash (Skin and subcutaneous tissue disorders) | 4/111 | 5/90 | 3/111 | 4/99 | 14/268 | 16/274
Hypertension (Vascular disorders) | 5/111 | 0/90 | 3/111 | 6/99 | 22/268 | 17/274
Dyspepsia (Gastrointestinal disorders) | 1/111 | 0/90 | 3/111 | 5/99 | 0/268 | 0/274
Infections and Infestations (General disorders) | 47/111 | 33/90 | 49/111 | 42/99 | 0/268 | 0/274
Gastroenteritis (General disorders) | 7/111 | 1/90 | 1/111 | 1/99 | 0/268 | 0/274
Lower respiratory tract infection (General disorders) | 2/111 | 1/90 | 4/111 | 5/99 | 0/268 | 0/274
Rhinitis (General disorders) | 2/111 | 2/90 | 6/111 | 1/99 | 0/268 | 0/274
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 13/111 | 11/90 | 15/111 | 9/99 | 0/268 | 0/274
Alanine aminotransferase increased (Investigations) | 5/111 | 7/90 | 2/111 | 1/99 | 0/268 | 0/274
Back pain (Musculoskeletal and connective tissue disorders) | 2/111 | 3/90 | 4/111 | 6/99 | 0/268 | 0/274
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/111 | 7/90 | 2/111 | 3/99 | 0/268 | 0/274
Depression (Psychiatric disorders) | 1/111 | 5/90 | 0/111 | 0/99 | 0/268 | 0/274

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.